CLINICAL TRIAL: NCT00622245
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, and Active Referenced Study of Lu AA34893 to Evaluate the Efficacy and Safety of Three Doses Lu AA34893 in the Treatment of Depression in Patients With Bipolar I or II Disorder
Brief Title: Efficacy and Safety of Lu AA34893 in Patients With Bipolar Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Human metabolite not yet covered sufficiently by nonclinical data
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12022A; 2007-002551-17 (EudraCT Number)
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Depression in Patients With Bipolar Disorder
Keywords: Depression; Bipolar disorder; Placebo-controlled; Double-blind; Multicenter; Clinical study; Mania
MeSH Terms: conditions — Depression; Bipolar Disorder; Mania | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lu AA34893: 4 mg (Experimental)
  Interventions: Drug: Lu AA34893
- Lu AA34893: 12 mg (Experimental)
  Interventions: Drug: Lu AA34893
- Lu AA34893: 18 mg (Experimental)
  Interventions: Drug: Lu AA34893
- Quetiapine fumarate (Other): Active reference 300 mg
  Interventions: Drug: Quetiapine fumarate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AA34893 — per oral doses, divided in twice daily administrations as capsules, during 12 weeks, followed by a one-week tapering period
  Arms: Lu AA34893: 12 mg; Lu AA34893: 18 mg; Lu AA34893: 4 mg
Drug: Quetiapine fumarate — per oral, once daily, during 12 weeks, followed by a one-week tapering period
  Arms: Quetiapine fumarate
Drug: Placebo — per oral doses, twice daily as capsules during 13 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of different doses of Lu AA34893 in the treatment of depression in patients with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder is a common lifelong psychiatric disorder. It is characterized by recurrent mood swings with manic or hypomanic episodes alternated with depressive episodes of longer duration. Patients spend more time in depression than in (hypo)mania over their life time. The medical need for the patient is to remain symptom-free for as long a period as possible. A reduction both in severity of depression and mania, and in frequency of cycling, is the aim.

Although there are many treatments for bipolar disorder, few are approved, and they have limitations in their use due to safety and tolerability issues. Recommendations exist to use mood stabilisers, antipsychotics or a combination thereof with or without antidepressants and the polypharmacy employed in many cases is a reason for concern. There is a major medical need for more effective treatments in monotherapy with a reduced potential for adverse effects. This study evaluates the efficacy and safety of the new drug, Lu AA34893, in treatment of depression in patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive episode of bipolar I or bipolar II disorder, according to DSM-IV TR
* Moderate to severe depression
* History of at least one documented mania or hypomania episode
* Absence of current mania or hypomania

Exclusion Criteria:

* Any current psychiatric disorder other than bipolar disorder defined in the DSM-IV TR
* Any substance disorder with the previous 6 months
* Use of any psychoactive medication (including mood stabilizers) within 2 weeks before randomisation and during the study
* ECT within 6 months before the study
* Female of childbearing potential and not using adequate contraception

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms as measured by the change from baseline in total MADRS score | 8 weeks

SECONDARY OUTCOMES:
HAM-D, CGI-BP, responders and remitters, BDI-II, HAM-A, safety parameters YMRS, AIMS, BARS, SAS, adverse events, clinical laboratory, ECG, physical examinations | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (50):
- Australia (3):
  - AU001, Brisbane
  - AU003, Dandenong
  - AU002, Malvern
- Austria (3):
  - AT002, Vienna
  - AT001, Vienna
  - AT003, Vienna
- Belgium (3):
  - BE004, Brussels
  - BE003, Charleroi
  - BE002, Diest
- BG004, Stara Zagora, Bulgaria
- Canada (3):
  - CA303, London
  - CA301, Montreal
  - CA302, Orléans
- France (4):
  - FR001, Clermont-Ferrand
  - FR007, Orvault
  - FR004, Paris
  - FR002, Sartrouville
- Germany (3):
  - DE004, Berlin
  - DE003, Bochum
  - DE002, Gelsenkirchen
- Lithuania (5):
  - LT005, Kaunas
  - LT003, Kaunas Region
  - LT004, Klaipėda
  - LT001, Vilnius
  - LT002, Vilnius
- Malaysia (3):
  - MY004, Klang
  - MY005, Kota Kinabalu
  - MY002, Kuala Lumpur
- Philippines (3):
  - PH002, Las Piñas
  - PH003, Mandaluyong
  - PH001, Mandaue City
- PL002, Gdansk, Poland
- Romania (4):
  - RO001, Arad
  - RO002, Bucharest
  - RO003, Cluj-Napoca
  - RO005, Craiova
- Slovakia (2):
  - SK001, Bratislava
  - SK002, Prešov
- South Korea (4):
  - KR004, Inchon
  - KR003, Jeonju
  - KR005, Kyunggi-do
  - KR002, Seoul
- Sweden (5):
  - SE006, Halmstad
  - SE003, Lund
  - SE005, Malmo
  - SE002, Sollentuna
  - SE001, Stockholm
- TW002, Taichung, Taiwan
- UA003, Lviv, Ukraine
- GB001, Oxford, United Kingdom